CLINICAL TRIAL: NCT06598423
Title: Pilot Test of a Novel Wavelength-Based Method to Control Childhood Myopia
Brief Title: Wavelength Intervention for Nearsighted Kids
Acronym: WINK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Safal Khanal, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 300013348; R21EY036536 (NIH)
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Myopia
Keywords: Childhood Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: The investigators plan to conduct a randomized controlled trial of specialized soft contact lenses for the treatment of myopia. Children will be randomized 1:1 to wearing a single type of soft contact lens or two types of soft contact lenses at alternate times daily for one year.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group A (Experimental): Children who are randomized to this group will wear one type of daily use, daily disposable, single-vision soft contact lens for at least four hours starting in the afternoon (after school) and another type of daily use, daily disposable, single-vision soft contact lens for the remainder of the time daily for one year.
  Interventions: Device: Specialized soft contact lens 1
- Control group (Sham Comparator): Children who are randomized to this group will wear daily use, daily disposable, single-vision soft contact lenses full time for one year. Contact lenses will be worn for a minimum of 10 hours per day.
  Interventions: Device: Specialized soft contact lens 2

INTERVENTIONS:
Device: Specialized soft contact lens 1 — These are daily-wear, daily-replacement lenses. They are identical to specialized soft contact lens 2 in material, comfort, and lens geometry. They differ only in their spectral profile.
  Arms: Group A
Device: Specialized soft contact lens 2 — These are daily-wear, daily-replacement lenses. They are identical to specialized soft contact lens 1 in material, comfort, and lens geometry. They differ only in their spectral profile.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to learn if daily brief periods of specialized soft contact lens wear work to slow the progression of nearsightedness in children. Additionally, the study will learn about the compliance and safety of specialized soft contact lens wear in children. The main questions it aims to answer are:

Does wearing specialized soft contact lenses daily slow myopia progression and axial elongation? What visual/ocular problems do participants have when wearing specialized soft contact lenses? Researchers will compare two soft contact lenses to see if specialized soft contact lens wear works to treat childhood myopia progression.

Participants will

1. Wear either a single type of soft contact lens or two types of soft contact lenses at alternate times daily full time in both eyes for one year.
2. Visit the clinic at 2 weeks, 1 month, 3 months, 6 months, and 12 months for checkups and tests
3. Keep a diary of the lens-wearing times.

DETAILED DESCRIPTION:
Myopia (nearsightedness) is a major public health concern. The prevalence of myopia continues to rise globally, including in the United States. Myopia develops when the eye grows excessively long for its optics, producing out-of-focus images of distant objects on the retina. Blurry distant vision in myopia can be easily corrected by traditional optical and surgical means. However, these methods do nothing to slow myopia-associated excessive axial elongation of the eye which is a major risk factor for several sight-threatening ocular pathologies, such as myopia maculopathy and retinal detachment later in life. Interventions to slow axial elongation and therefore myopia will have a significant public health benefit.

This randomized controlled clinical trial will test the efficacy of wearing specialized soft contact lenses in slowing the progression of myopia in children. In this pilot trial, children with myopia will wear daily use, daily disposable, single-vision soft contact lenses in both eyes for one year. One group will wear a single type of soft contact lens full-time daily whereas the other group will wear two types of soft contact lenses daily at alternate times. The two lenses are identical in material, comfort, and lens geometry and different only in their spectral profile.

ELIGIBILITY:
Inclusion Criteria:

* Spherical component of refractive error in primary meridian between -0.75 and -5.00 D
* Less than 1.00 D of astigmatism or anisometropia
* History of soft contact lens wear for at least a week
* Best-corrected visual acuity of 20/25 (+0.10 logMAR) or better in each eye
* Willingness to wear the lenses for a minimum of 10 hours/day, at least six days a week for the duration of the study

Exclusion Criteria:

* Subjects receiving myopia control treatments within the past six months
* History of premature (less than 3.3 lb) or preterm birth (earlier than 30 weeks)
* Current history of using systemic or ocular medications (including artificial tears) that may affect contact lens wear, tear film health, refractive state, pupillary response or accommodative function
* History of ocular or systemic diseases, including those that may affect refractive development
* Known allergy to fluorescein, benoxinate, proparacaine, or tropicamide
* Contact lens contraindications (e.g., giant papillary keratoconjunctivitis)
* Corneal disorders (e.g., hypoesthesia, keratoconus)
* Strabismus at distance or near with distance glasses or contact lenses
* Subjects exhibiting poor personal hygiene that may affect the compliance of contact lens wear.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in cycloplegic spherical equivalent refractive error | Baseline and 12 months
  Cycloplegic autorefraction measurements will be recorded using the WAM 5500 autorefractor in both eyes at baseline and follow-up visits. A set of 10 spherical equivalent measures will be obtained in each eye and later averaged to obtain the eye's final refractive error.
Change in axial length | Baseline and 12 months
  Ocular component dimensions, including axial length, will be recorded using the Haag-Streit LenStar LS900 based on low-coherence interferometry. A set of five measurements in primary gaze in each eye will be averaged to obtain the final dimension of the ocular components.

SECONDARY OUTCOMES:
Change in choroidal thickness | Baseline and 12 months
  Subjects will have cross-sectional chorio-retinal images taken in each eye using a high resolution scan centered on the fovea in the enhanced depth imaging mode. After the scanning is complete, images will be exported in original resolution for offline processing in MATLAB using custom software that will segment layers and automatically measure choroidal thickness at various regions (subfoveal, central, parafoveal, peripheral) as the distance between the retinal pigment epithelium/choroid interface and the choroidoscleral interface.
Change in visual acuity | Baseline and 12 months
  High-contrast distance visual acuity (VA) will be measured at 4 m with ETDRS Charts and near VA will be measured at 40 cm with Near Point Flip Charts. Low-contrast VA will be measured using 10% contrast Bailey Lovey charts. Monocular VA will be recorded in logMAR to the nearest letter on charts standardized to a luminance of 85 cd/m2.
Change in accommodative response | Baseline and 12 months
  A Grand Seiko autorefractor WAM 5500 will be used to measure accommodative response while fixating at 20/100 letters at 40 and 25 cm.

CONTACTS AND LOCATIONS:
Overall Officials: Safal Khanal, OD, PhD, Principal Investigator — Unversity of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham School of Optometry, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in myopia. Data will be coded, with no PHI included. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact skhanal@uab.edu.

REFERENCES:
- [Background] Khanal S, Norton TT, Gawne TJ. Amber light treatment produces hyperopia in tree shrews. Ophthalmic Physiol Opt. 2021 Sep;41(5):1076-1086. doi: 10.1111/opo.12853. Epub 2021 Aug 11. PMID 34382245
- [Background] Gawne TJ, Grytz R, Norton TT. How chromatic cues can guide human eye growth to achieve good focus. J Vis. 2021 May 3;21(5):11. doi: 10.1167/jov.21.5.11. PMID 33984119
- [Background] Gawne TJ, She Z, Khanal S. Human trichromacy and refractive development. Vision Res. 2025 Sep;234:108632. doi: 10.1016/j.visres.2025.108632. Epub 2025 Jun 9. PMID 40494187